CLINICAL TRIAL: NCT04151693
Title: Health Psychological Group Rehabilitation for Patients With Chronic Fatigue Syndrome (ME/CFS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: TheWellbeing Services County of Pirkanmaa (Unknown); Charite-Institute of Medical Immunology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D/1964/13.00.00.00/2019 Q 028
Record Dates: First submitted 2019-09-24; First posted 2019-11-05 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Psychological Adaptation; Cognitive Change; Adaptive Behavior; Functioning
Keywords: Psychological intervention; Cognitive Behavioral Therapy (CBT); Accept and Commitment Therapy (ACT); Cognitive functioning; Fatigue; Autonomic nervous system; Autonomic nervous system ganglio antibodies; Deep breathing; Relaxation; Health care system; Agency; Health psychology; Pacing
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Research group, 35-40 participants (8 sessions in 4 months) Control group (health and lifestyle counselling), 35-40 participants (6 sessions in 3 months)
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Research group ME/CFS (Experimental): Health Psychological Group Rehabilitation for Patients With Chronic Fatigue Syndrome (ME/CFS)
  8 sessions in 4 months. n=35-40 patients
  ME/CFS -Current knowledge Smart goals Stress management in every day life Pacing Psychological effects of illness and adaptation Coping strategies Emotional support Focus on autonomic nervous system (hyperarousal, cognitive disabilities) Focus on health
  Interventions: Behavioral: Health Psychological Group Rehabilitation for Patients With Chronic Fatigue Syndrome (ME/CFS)
- Control group ME/CFS (Experimental): Control group
  6 sessions in 3 months n=35-40 patients
  Health, lifestyle and wellbeing counselling (sleep, nutrition, activities in daily life)
  Interventions: Behavioral: Health Psychological Group Rehabilitation for Patients With Chronic Fatigue Syndrome (ME/CFS)

INTERVENTIONS:
Behavioral: Health Psychological Group Rehabilitation for Patients With Chronic Fatigue Syndrome (ME/CFS) — Adaptation (support own agency), rehabilitation and improvement of functional capacity.

SUMMARY:
Chronic fatigue syndrome (ME/CFS) is a severe medical condition. It is characterized by long term fatique and other persisted symptoms, such as a cognitive disabilities and orthostatic intolerance. Symptoms limit a persons ability to carry out ordinary daily activities. In ICD- 10, disease is known as G93.3, postviral fatigue syndrome.

The purpose of this research (doctoral study) is to produce a health psychological group intervention for patients with ME/CFS.

Research protocol: 70-80 patients with diagnosis G 93.3. Psychological and psychiatric evaluation for patients (SCID I and parts from SCID II). Depression diagnosis is allowed (on remission). Medication for depression is also allowed. Measurements for ortostatic intolerance (Somnotouch nimbTM) and laboratory measurements: complete blood count, CRP, alkaline phosphatase, GT, ALAT, CK, bilirubin, kidney and thyroid (TSH, T4V) function tests, serum ferritin, glucose, electrolytes and daily urine sodium excretion.

Autonomic nervous system ganglio antibodies: Anti-AT1R- Antibodies, Anti- ETAR- Antibodies, anti alpha-1 adrenergic Receptor Antibodies, anti alpha 2 adrenergic Receptor Antibodies, anti beta-1 adrenergic Receptor Antibodies, anti beta-2-adrenergic Receptor Antibodies, anti- Muscarinic Cholinergic Receptor 1 (M1)- Antibodies, anti- Muscarinic Cholinergic Receptor 2 (M2)- Antibodies, anti- Muscarinic Cholinergic Receptor 3 (M3)- Antibodies, anti- Muscarinic Cholinergic Receptor 4 (M4)- Antibodies, anti- Muscarinic Cholinergic Receptor 5 (M5)- Antibodies.

DETAILED DESCRIPTION:
Testing and inventories before rehabilitation/ at the end of the rehabilitation and 3 months follow-up.

1. ME/CFS patients modalities of agency.The study includes five patients with chronic fatigue syndrome and examines their modalities of agency. A special focus is on the effects of the health care system on the patients' agency.The research is qualitative, the data was analyzed using theory-driven content analysis.
2. The study explores the experiences of Health Psychological group rehabilitation for patients with ME/CFS. The aim is to better overall functioning and management of illness through goal-oriented work, dealing emotions with the crisis of the illness, adopting, and implementing healthy lifestyle choices. The study is qualitative (n=10) using content analysis.
3. Randomized controlled research. n=70. Treatment/research group n=35. Control- group (35) participates on health counselling (6 sessions). Research question: is health psychological group rehabilitation clinically statistically significant. Comparison is between research- and control groups but also between patients who are diagnosed 93.3, having also objective impairment in cognitive functions or orthostatic intolerance, comparing to patients only diagnosed on G93.3.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic fatigue syndrome, G 93.3
* Must be able to sit two hours and do homework tasks
* Must be motivated to co-operate with other patients
* Goal oritentation
* Have an interest to learn health psychological approach and willingness to participate rehabilitation

Exclusion Criteria (diseases without treatment/ acute phase):

* hypothyroidism
* sleep apnea or narcolepsy
* major depressive disorders, bipolar affective disorders, schizophrenia
* eating disorders
* cancer
* autoimmune disease
* hormonal disorders
* subacute infections
* obesity
* alcohol or substance abuse
* vitamin D deficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
WHODAS 22.0 (World Health Organization Disability Assessment Schedule) 2.0. | Before intervention and change immediately after the intervention and 3 months follow up
  36 questions, scale 0-5 (not difficult at all-very difficult) Subscales: 1)communication with other people 2) Mobility/ movement in everyday activities 3)Daily functions and taking care of oneself 4) Relationships 5) Daily routines 6) Disabilities in last 30 days 7)Participating on community
COMPASS31 | Before intervention and change immediately after the intervention and 3 months follow up
  Autonomic nervous system/ neurological symptoms, inventory,31 questions. Subscales: different neurological symptoms, scales from 0-1 to 0-7. Score is reported on subscales.

SECONDARY OUTCOMES:
HADS (Hospital Anxiety and Depression Scale) | Before intervention and change immediately after the intervention and 3 months follow up
  Depression and anxiety, inventory,14 questions, scale 0-3. Total score is reported (0-7:normal- 8-10:borderline-11-21:abnormal)
SOC-14 (Sense Of Coherence) | Before intervention and change immediately after the intervention and 3 months follow up
  Sense of coherence, inventory, 14 questions, scale 0-7. Total score is reported/ scores are reported on subscales: (comprehensibility, manageability, meaningfulness)
FSS (Fatigue severity scale) | Before intervention and change immediately after the intervention and 3 months follow up
  Fatigue severity scale,9 questions, scale 0-7 (I strongly disagree- I strongly agree) total score is reported.
PHQ-4 (patient health questionnaire) | Before intervention and change immediately after the intervention and 3 months follow up
  Depression and anxiety, inventory, 4 guestions. Subscales: anxiety and depression. Total score is reported ( 0-1 none,3-5 mild, 6-8 moderate, 10-12 severe)

CONTACTS AND LOCATIONS:
Overall Officials: Tuomo Nieminen, Study Chair — Päijät- Häme Joint Authority for Health and Wellbeing
Locations (1):
- Päijät Häme Central Hospital, Lahti, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keurulainen M, Holma J, Wallenius E, Pankalainen M, Hintikka J, Partinen M. 'I became more aware of my actions'-A qualitative longitudinal study of a health psychological group intervention for patients with myalgic encephalomyelitis/chronic fatigue syndrome. Health Expect. 2023 Dec;26(6):2312-2324. doi: 10.1111/hex.13833. Epub 2023 Aug 1. PMID 37528544